CLINICAL TRIAL: NCT01961206
Title: Community-Onset Bacteremia Due to Extended-Spectrum β-Lactamase (ESBL)Producing Escherichia Coli or Klebsiella Pneumoniae in China: Prevalence, Risk Factors and Prognosis
Brief Title: Community-Onset Bacteremia Due to ESBL Producing E.Coli or K.Pneumoniae in China: Prevalence, Risk Factors and Prognosis
Status: Completed | Type: Observational
Sponsor: Jian-cang Zhou M.D. (Other)
Responsible Party: Sponsor-Investigator, Jian-cang Zhou M.D., Dr., Sir Run Run Shaw Hospital
Organization: Sir Run Run Shaw Hospital (Other)
Other Study IDs: SRRSH-ESBL01
Record Dates: First submitted 2013-09-30; First posted 2013-10-11 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Community Acquired Infection
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacterial strains
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Patients: Case Patients with Community-Onset Bacteremia Due toESBL producing E.coli or K.pneumoniae
  Interventions: Other: bacteremia caused by ESBL producing E.coli or K.pneumoniae
- control group: bacteremia caused by ESBL producing E.coli or K.pneumoniae

INTERVENTIONS:
Other: bacteremia caused by ESBL producing E.coli or K.pneumoniae — community-onset bacteremia caused by ESBL producing E.coli or K.pneumoniae
  Groups: Case Patients

SUMMARY:
Escherichia coli is the leading cause of community-onset gram-negative bloodstream infections. There has been a dramatic increase in the prevalence of extended-spectrum b-lactamases producing E. coli and K.pneumoniae in the community, which was considered to be exclusively a nosocomial pathogen in recent years. As a result, the treatment options for community-onset infections due to ESBL-producing E. coli or K.pneumoniae are limited and the initial empirical therapy is often ineffective and associated with increased mortality. Although there were some reports of the risk factors of community-onset ESBL producing E. coli in Spain, Korea, and Canada, few empirical data were available about China. Therefore, the investigators aim was to investigate the epidemiology, risk factors, and the hospital outcomes for patients with community-onset bacteremia caused by ESBL producing E. coli or K.pneumoniae in China.

DETAILED DESCRIPTION:
Eligibility criteria:

1. Inclusion criteria:Blood cultures demonstrated E.coli or K.pneumoniae among nonhospitalized patients or within 48 h after hospitalization.
2. Exclusion criteria:Patients with hospitalization in the past 1 month.

Outcome measures:

1. Risk factors for community-onset bacteremia due to ESBL producing E. coli or K.pneumoniae
2. Microbial and clinical efficacy of commonly used antibiotics for community-onset bacteremia due to ESBL producing E. coli or K.pneumoniae

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* community-onset bacteremia

Exclusion Criteria:

* recent hospitalization within one month in any hospital

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients visited any of the 28 particitant hospitals during the study period were screened. Patients with community-onset bacteremia caused by E.coli or K. pneumoniae and without a recent hospitalization in any hospital will be included
Sampling Method: Non-Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Risk factors for community-onset bacteremia caused by ESBL producing E.coli or K.pneumoniae | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song YU, M.D, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Rodriguez-Bano J, Picon E, Gijon P, Hernandez JR, Ruiz M, Pena C, Almela M, Almirante B, Grill F, Colomina J, Gimenez M, Oliver A, Horcajada JP, Navarro G, Coloma A, Pascual A; Spanish Network for Research in Infectious Diseases (REIPI). Community-onset bacteremia due to extended-spectrum beta-lactamase-producing Escherichia coli: risk factors and prognosis. Clin Infect Dis. 2010 Jan 1;50(1):40-8. doi: 10.1086/649537. PMID 19995215
- [Result] Apisarnthanarak A, Kiratisin P, Mundy LM. Predictors of mortality from community-onset bloodstream infections due to extended-spectrum beta-lactamase-producing Escherichia coli and Klebsiella pneumoniae. Infect Control Hosp Epidemiol. 2008 Jul;29(7):671-4. doi: 10.1086/588082. PMID 18624669
- [Derived] Quan J, Zhao D, Liu L, Chen Y, Zhou J, Jiang Y, Du X, Zhou Z, Akova M, Yu Y. High prevalence of ESBL-producing Escherichia coli and Klebsiella pneumoniae in community-onset bloodstream infections in China. J Antimicrob Chemother. 2017 Jan;72(1):273-280. doi: 10.1093/jac/dkw372. Epub 2016 Sep 13. PMID 27624571